CLINICAL TRIAL: NCT07251816
Title: Neural Bases of Motivation
Acronym: MOTIVACTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 69HCL25_0205; 2025-A00984-45 (Other: ID-RCB)
Record Dates: First submitted 2025-09-01; First posted 2025-11-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Motivation; Action
Keywords: Healthy volunteers; Motivation; Apathy; Decision-making; Effort processing
MeSH Terms: conditions — Lethargy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Experiments 1 to 5 require randomization of the stimulation conditions within each participant, either across sessions (in experiments 1, 2, 3, and 4) or across blocks of trials (in experiment 5).
  Only the principal investigator have the list of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Experiment 1 (Experimental): First, participant will undergo a structural magnetic resonance imaging (MRI). Then, participant will come to the scanner for 3 sessions. In each of the three sessions, participant will first perform the effort-based decision-making task in the functional (f)MRI scanner to establish baseline measures of decision behavior and connectivity. Following this, cortico-cortical paired associative stimulation will be applied using one of three conditions:
  1. the supplementary motor area will be stimulated first, followed by the motor cortex.
  2. the motor cortex will be stimulated first, followed by the supplementary motor area.
  3. control stimulation, where the supplementary motor area will be stimulated first, followed by the motor cortex with a minimal 1 ms delay, which will not modulate effective connectivity.
  After stimulation, participant will again perform the effort-based decision-making task in the fMRI scanner.
  Interventions: Procedure: Cortico-cortical paired-associative stimulation (ccPAS); Procedure: MRI; Procedure: Pupillometry; Behavioral: Neuropsychological scales
- Experiment 2 (Experimental): First, participant will undergo a structural MRI scan. Then, participant will come for three sessions. In each session, participants will begin by performing the effort-based decision-making task while their baseline behavioral and neural activity is recorded using electroencephalography (EEG). Following this initial task, bifocal transcranial alternating current stimulation (tACS) will be applied under one of three conditions:
  1. real, in-phase stimulation to synchronize oscillations between the supplementary motor area and motor cortex;
  2. real, in-phase stimulation to synchronize oscillations between the orbitofrontal cortex and motor cortex;
  3. control stimulation, where oscillations between the supplementary motor area and the motor cortex are applied in antiphase.
  Participant will perform the decision-making task during the stimulation. After the stimulation, participant will repeat the decision-making task with EEG recording.
  Interventions: Procedure: Bifocal transcranial alternating current stimulation (tACS); Procedure: MRI; Procedure: Pupillometry; Behavioral: Neuropsychological scales; Procedure: EEG
- Experiment 3 (Experimental): First, participant will undergo a structural MRI scan. Then, participants will come to the lab to record electroencephalography (EEG) for three sessions. In each session, participant will begin by performing the effort-based decision-making task with EEG recording. Following this initial task, combined oscillatory magnetic stimulation and temporal interference stimulation will be applied under one of three conditions:
  1. real oscillatory magnetic stimulation combined with real temporal interference stimulation;
  2. control oscillatory magnetic stimulation (using a control coil, making the same noise as a real stimulation) combined with real temporal interference stimulation;
  3. both control oscillatory magnetic stimulation and a control temporal interference stimulation as a control condition.
  Participant will perform the decision-making task during stimulation. After the stimulation, participant will repeat the decision-making task with EEG recording.
  Interventions: Procedure: Combining transcranial temporal interference stimulation (tTIS) and oscillatory TMS; Procedure: MRI; Procedure: Pupillometry; Behavioral: Neuropsychological scales; Procedure: EEG
- Experiment 4 (Experimental): Participant will come to the MRI facilities for three sessions. In each session, participants will begin by performing the effort-based decision-making task while their baseline behavioral and neural activity is recorded using fMRI. Following this initial task, transcranial direct current stimulation will be applied under one of three conditions:
  1. real anodal stimulation,
  2. real cathodal stimulation,
  3. control stimulation. Participant will perform the decision-making task during stimulation. Further, stimulation will be realized in the scanner using an MRI-compatible set-up, to directly measured the changes in neural activity induced by the stimulation.
  After the stimulation, participants will repeat the decision-making task with fMRI recording.
  Interventions: Procedure: Transcranial direct current stimulation (tDCS); Procedure: MRI; Procedure: Pupillometry; Behavioral: Neuropsychological scales
- Experiment 5 (Experimental): Participant will come to the MRI facilities for one experimental session. In this single session, participant will first perform the task while transcutaneous vagal nerve stimulation will be applied under one of two conditions in separate blocks of trials:
  1. real stimulation, aimed at modulating the activity of the locus coeruleus and influencing the noradrenergic system;
  2. control stimulation, which serves as a control to account for non-specific effects of the procedure.
  During the stimulation, participant will continue performing the decision-making task.
  Interventions: Procedure: Transcutaneous vagal nerve stimulation (tVNS); Procedure: MRI; Procedure: Pupillometry; Behavioral: Neuropsychological scales
- Preparatory experiment 1 (Experimental): First, each participant will undergo a structural magnetic resonance imaging session at the CERMEP. The acquired data will be used for neuro-navigation, ensuring precise targeting of brain regions during the paired-pulse stimulation procedure.
  Then, participants will perform the effort-based decision-making task while paired-pulse stimulation is applied during the decision-making period. The stimulation will target circuits connecting the supplementary motor area and the motor cortex. Test pulses will be delivered to the motor cortex, either alone or preceded by a conditioning pulse to the supplementary motor area. These conditioned and unconditioned stimulations will occur at random intervals during the decision-making phase of the task. Motor-evoked potentials will be recorded with surface electromyography throughout the decision-making period.
  Interventions: Procedure: Cortico-cortical paired-associative stimulation (ccPAS); Procedure: MRI; Procedure: Pupillometry; Behavioral: Neuropsychological scales
- Preparatory experiment 2 (Experimental): First, participants will perform the effort-based decision-making task while MEG is used to record neural oscillatory activity (one session). This recording will take place at the MEG facility of the CERMEP, ensuring high temporal and spatial precision in capturing brain dynamics during task performance.
  Then, each of the participants will undergo a structural MRI scan that will be used to improve source localization during MEG data processing.
  Interventions: Procedure: MRI; Procedure: MEG; Procedure: Pupillometry; Behavioral: Neuropsychological scales

INTERVENTIONS:
Procedure: Cortico-cortical paired-associative stimulation (ccPAS) — Transcranial magnetic stimulation (TMS)
  Arms: Experiment 1; Preparatory experiment 1
Procedure: Bifocal transcranial alternating current stimulation (tACS) — Transcranial electrical stimulation (tES)
  Arms: Experiment 2
Procedure: Combining transcranial temporal interference stimulation (tTIS) and oscillatory TMS — Transcranial electrical stimulation and transcranial magnetic stimulation
  Arms: Experiment 3
Procedure: Transcranial direct current stimulation (tDCS) — Transcranial electrical stimulation
  Arms: Experiment 4
Procedure: Transcutaneous vagal nerve stimulation (tVNS) — Transcutaneous vagal nerve stimulation (tVNS)
  Arms: Experiment 5
Procedure: MRI — Magnetic Resonance Imaging
Procedure: MEG — Magnetoencephalography
  Arms: Preparatory experiment 2
Procedure: Pupillometry — Measurement and analysis of changes in pupil diameter over time, providing a non-invasive and straightforward method to investigate physiological and psychological processes. Using an eye tracker or pupillometer equipped with infrared cameras, pupil size is measured with high precision and temporal resolution. Pupil responses serve as a proxy for effort invigoration and are linked to multiple neuromodulatory systems, including the noradrenergic system. Recordings will be conducted throughout both experiments, with participants instructed to minimize movements and blinking to ensure data quality.
Behavioral: Neuropsychological scales — Different neuropsychological scales will be administered to assess various psychological and behavioral dimensions relevant to the study, such as: the Apathy Evaluation Scale (AES): To evaluate levels of apathy ; the Depression Anxiety Stress Scale (DASS): To assess depression, anxiety, and stress ; and the Snaith-Hamilton Pleasure Scale (SHAPS): To evaluate the inability to experience pleasure.
Procedure: EEG — Electroencephalography
  Arms: Experiment 2; Experiment 3

SUMMARY:
Effort-based decisions are essential in daily life but strongly impaired in apathy across various brain disorders. Now, significant research to unveil the neural causes of apathy is needed. A crucial corollary to this is the need to identify the brain network and neural mechanisms underlying effort-based decisions.

A fronto-striatal network and the noradrenergic system are involved in effort-based decision-making and apathy. Further, motor cortical structures may play a role in effort-based decision-making. However, the role of circuits connecting the fronto-striatal network and the noradrenergic system to the motor structures has been disregarded so far.

Non-invasive brain stimulation methods provide a unique and safe means to test the causal role of connectivity changes between fronto-subcortical and motor structures in effort-based decision-making.

It's now necessary to have an integrative, connectionnist framework to uncover the causal role of connectivity changes between fronto-subcortical and motor structures in effort-based decision-making.

The overarching goal of the present research protocol is to establish an integrative framework testing the causal role of connectivity within recurrent, bidirectional circuits between fronto-subcortical circuits and motor structures in effort-based decision-making. To achieve this overarching goal, investigators will quantifiy the causal role of effective connectivity and oscillatory synchrony in these circuits on effort-related behavior using a non-invasive brain stimulation strategy. Further, a secondary aim is to identify potential non-invasive brain stimulation methods that could increase engagement in effortful behavior, paving the way for translational clinical applications in the context of apathy.

The investigators hypothesize that effort-based decision-making in healthy subjects is governed by bidirectional interactions between fronto-subcortical circuits and motor structures such as the primary motor cortex, mediated by oscillatory synchrony in specific frequency bands (e.g., theta and gamma bands). Accordingly, they hypothesize that transient, non-invasive modulation of connectivity and oscillatory synchrony between these structures in healthy human subjects will directly modulate their decision to engage in effort. Specifically, five experiments will use complementary approaches to test the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged between 18 and 40 years
* Participants without confounding factors such as neural alterations related to neurological pathology, whether neurodegenerative (e.g., Alzheimer, Parkinson, Huntington, multiple sclerosis, amyotrophic lateral sclerosis), motor (e.g., dystonia, essential tremors, cerebellar syndrome), traumatic (e.g., traumatic brain injury, medulla lesion) or psychiatric pathologies, whether mood disorders (e.g., depression, bipolarity), anxious troubles (e.g., obsessional compulsive disorder, post-traumatic stress disorder), psychotic (e.g., schizophrenia, delusion), substance-related (e.g., alcool, drug or medicine addiction), food-related (e.g., anorexia, bulimia), neurodevelopmental (e.g., autism, attention-deficit with hyperactivity disorder) or personality (e.g., borderline personality disorder, antisocial personality disorder, obsessive-compulsive disorder).
* Participants affiliated with a compulsory social security scheme.

Exclusion Criteria:

* Persons deprived of liberty by judicial or administrative decisions.
* Pregnant women, women in labor or breastfeeding women
* Persons admitted to a health or social institution for purposes other than research.
* Adults under legal protection measures (e.g., guardianship or curatorship).
* Participation in other interventional research with an ongoing non-inclusion period.
* Neurological or psychiatric disorders.
* Use of tricyclic antidepressants (amitriptyline, clomipramine, imipramine, nortriptyline), neuroleptics (chlorpromazine, haloperidol, risperidone, olanzapine, quetiapine), or recreational drugs within the past 48 hours.
* Regular use of recreational drugs.
* Sleep deprivation (< 5 hours regularly over the last 3 months)
* Left-handedness or ambidexterity.
* Physical injuries impacting motor tasks.
* Presence of metal implants in the head (excluding oral fillings).
* Presence of implanted medical devices (e.g., pacemaker).
* Presence of metallic injuries in the eyes.
* Claustrophobia.
* Piercings incompatible with MRI procedures.
* Contraindication to MRI
* Persons who refused to be informed of eventual medical anomalies discovered by the MRI
* Personal or family history (first-degree relatives) of epilepsy or seizures. Severe and/or frequent headaches (only for participants receiving transcranial magnetic stimulation, e.g preparatory experience 1 and experience 1)
* Baldness impeding electrode placement (only for participants receiving transcranial electrical stimulation and EEG measurements, e.g experiments 2, 3 and 4)
* Facial or ear pain and/or recent ear trauma (only for participants receiving transcutaneous vagal nerve stimulation, e.g experiment 5)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Acceptance rates (from 0 to 100 % of acceptance) for behavioral outcomes. Connectivity and oscillatory changes for neural activity | Up to 6 months
  Acceptance rate is the participant's willingness to engage in effortful tasks for rewards and reaction times measure the rapidity to approach or avoid the effort.
  Connectivity and oscillatory changes will be analyses with imaging data
Reaction times (in ms) for behavioral outcomes. Connectivity and oscillatory changes for neural activity | Up to 6 months
  Acceptance rate is the participant's willingness to engage in effortful tasks for rewards and reaction times measure the rapidity to approach or avoid the effort.
  Connectivity and oscillatory changes will be analyses with imaging data

SECONDARY OUTCOMES:
fMRI connectivity | Up to 6 months
  fMRI-measured effective connectivity between cerebral structures
EEG-measured synchrony | Up to 6 months
  Measured synchrony as frequency coherence between cortical structures

CONTACTS AND LOCATIONS:
Locations (1):
- Equipe ImpAct CRNL, INSERM U1028 CNRS UMR 5292, Bron, France